CLINICAL TRIAL: NCT05595681
Title: Effect of Mesenchymal Stem Cells on Healing of Foot Ulcers in Diabetes Patients. A Phase I Pilot Study.
Brief Title: Effect of Mesenchymal Stem Cells on Healing of Foot Ulcers in Diabetes Patients.
Acronym: STEMFOOT
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Difficulties in enrolling trial subjects within in- and exclusion criteria, despite the trial period having been extended several times.
Sponsor: Cell to Cure ApS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STEMFOOT Pilot study
Record Dates: First submitted 2022-09-23; First posted 2022-10-27 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Diabetic Foot Ulcer; Mesenchymal Stromal Cells
Keywords: Healing Ulcer; Complications
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Single center randomized open phase I clinical intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): 20 x 1000000 C2C_ASCs on top of standard care.
  Interventions: Drug: Adipose tissue derived mesenchymal stromal/stem cells (Cell2Cure®)
- Control group (No Intervention): Control group with standard care.

INTERVENTIONS:
Drug: Adipose tissue derived mesenchymal stromal/stem cells (Cell2Cure®) — The investigational product is a C2C_ASC cell product (Cell2Cure®, Cell2Cure ApS, Denmark).
  C2C_ASC is an advanced therapy investigational medicinal product (ATIMP) manufactured from abdominal adipose tissue derived mesenchymal stromal cells (ASC) from healthy donors. C2C_ASC is aseptically procured and manufactured according to tissue law and GMP by Cell2Cure ApS or Cardiology Stem Cell Center, Rigshospitalet, Copenhagen, Denmark, using manual isolation of cells from abdominal fat tissue, xeno-free cell expansion in automated closed bioreactor systems and cryopreservation of the final product.
  The active substance is the in vitro expanded ASCs. The final product, C2C_ASC, is provided as a cryopreserved suspension of 50 million ASCs per ml with a total volume of 1,3 ml per vial. The exipient is CryoStor10 (Biolife Solutions), holding 10% DMSO.
  Arms: Treatment group

SUMMARY:
The STEMFOOT Pilot Study is a single center randomized open phase I clinical intervention pilot trial with the aim of investigating the treatment effect of an allogenic adipose-derived mesenchymal stromal cell product (C2C_ASC) compared to conventional optimal treatment on healing and complications of foot ulcers in diabetes patients.

DETAILED DESCRIPTION:
The STEMFOOT Pilot Study will be performed at Copenhagen Diabetes Foot Center, Department of Endocrinology, Bispebjerg Hospital, Denmark. 30 adult patients with diabetes and foot ulcer will be enrolled and randomly assigned 1:1 to either C2C_ASC treatment on top of standard care (n=15) or control group with standard care (n=15).

C2C_ASC treatment: 1 ml containing 20 x 106 C2C_ASCs will be injected into the subcutaneous dermo-epidermal junction and homogenously around the wound (4 - 6 injections), but not directly within the index foot ulcer. The depth from the index wound border will be 0,5 - 1 cm into the subcutaneous tissue.

Standard care: Each treatment will be administered in the context of independently-managed standard of care, including (a) formal assessment of the ulcer and surrounding skin at each clinic review; (b) provision of any necessary off-loading, with detailed description of the type and assessment of its effectiveness; (c) debridement of the wound surface, which can be surgical (either in the clinic or in an operating room) or non-surgical; (d) selection of appropriate dressing products, ensuring a moist ulcer environment; (e) management of ulcer infection; (f) attention to nutrition and self-care; (g) optimization of glycemic and risk factor control; (h) revascularization when appropriate and (i) continued close observation with appropriate adjustment of management.

We hypothesize that in diabtes patients with foot ulcer, the time to healing is significantly shorter and more foot ulcers are completely healed at week 12 when treated with C2C_ASC on top of standard care compared to control.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes mellitus for at least 3 months.
* Age 40-75 years.
* A foot ulcer below the level of the malleoli, excluding ulcers confined to the digits or interdigital cleft. If more than one ulcer, the largest will be selected at screening as the index ulcer.
* Wound area after sharp debridement of ≥ 50 mm^2, but ≤1000 mm^2.

Exclusion Criteria:

* Signs of infection of the index ulcer.
* An ulcer where a probe investigation indicates ulcer depth to the underlying bone.
* Wound caused primarily by untreated vascular insufficiency, or where participants are primarily eligible for vascular intervention to promote wound healing.
* Wounds with an etiology not related to diabetes.
* Underlying osteomyelitis of the leg with the wound to be treated.
* Participants presenting with the clinical characteristics of cellulitis at the wound site (suppurative inflammation involving particularly the subcutaneous tissue, often mild erythema, tenderness, malaise, chills and fever).
* Surgery to lengthen achilles tendon on the leg with the wound to be treated 3 months prioer to signing the informed consent form.
* Necrosis, purulence, or sinus tracts that cannon be removed by debridement on foot to be treated.
* Toe blood pressure < 44 mmHg at the foot with the index ulcer.
* Dialysis or an estimated glomerular filtration rate (GFR) (based on serum creatinine) < 20 ml/min/1.73 m^2.
* Current treatment with cytotoxic drugs.
* Hospitalisation for a major cardiovascular event or procedure or revascularization surgery on a leg in the last 3 months or scheduled major cardiovascular intervention.
* Abuse of alcohol or drugs, or presence of any condition that in the Investigators opinion may lead to poor adherence to study protocol.
* Recent use (< 3 months) of an investigational drug or participation in interventional clinical foot ulcer-healing trial.
* Females capable of becoming pregnant must have a negative pregnancy test prior to transplantation. After inclusion, they must use contraceptives for 12 weeks following the given stem cell treatment. The pill, spirak, depot injection of progesterone, sub-dermal implantation, hormonal vaginal ring and transdermal patch regarded as safe contraceptives.
* Likely inability yo comply with the need for clinical visits because of planned activity.
* Mental incapacity, unwillingness, or language barrier precluding adequate understanding or cooperation.
* Unable to provide written and signed informed consent.
* Any clinically significant disease or disorder, except for conditions associated to the type 1 or 2 diabetes, which in the Investigator's opinion could interfere with the results of the trial.
* Active cancer or a history of cancer in the 5 years prior to signing the informed consent form (history of basal cell carcinoma is allowed).
* Life expectancy of less than 12 months.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2025-11-28 (Actual); Study Completion 2025-11-28 (Actual)

PRIMARY OUTCOMES:
Time to complete ulcer healing | 12 weeks
  Complete ulcer healing is defined as complete skin re-epithelialization without drainage or dressing requirements after removal of callus, confirmed at two consecutive study visits two weeks apart, and the time encountered as healed is the first of the two visits.

SECONDARY OUTCOMES:
Amount of index ulcers completely healed | 12 weeks
  Change in ulcer area at week 12

OTHER OUTCOMES:
Other endpoints | 12 weeks
  difference between groups of participant adverse events and serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Kastrup, Study Director — Cell to Cure ApS
Locations (1):
- Copenhagen Diabetes Foot Center (CODIF), Copenhagen, Denmark